CLINICAL TRIAL: NCT00799370
Title: Prospective Study on Postoperative Weight Bearing After Opening Wedge High Tibial Osteotomy (HTO): Early Weight Bearing Versus Delayed. Open Labelled Randomized Clinical Study
Brief Title: Randomized Control Trial on Postoperative Weight Bearing After High Tibial Osteotomy (HTO)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2007.477
Record Dates: First submitted 2008-11-25; First posted 2008-11-27 (Estimated); Last update posted 2019-05-28 (Actual); Status verified 2014-06

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteotomy; Weight bearing; Opening wedge
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Early weight bearing: immediate in postoperative
  Interventions: Procedure: Early weight bearing
- 2 (Experimental): Delayed weight bearing: 2 months after surgery
  Interventions: Procedure: Delayed weight bearing

INTERVENTIONS:
Procedure: Early weight bearing — Weight bearing performed immediately after surgery
  Arms: 1
Procedure: Delayed weight bearing — Weight bearing performed 2 months after surgery
  Arms: 2

SUMMARY:
The study analyzes the consequences of weight bearing after an HTO in a population of young patient with medial osteoarthritis (immediate weight bearing versus two month weight bearing). The two options are usually used so the protocol belongs to the intermediate care evaluation category.

The IKS (International Knee Society) score at one year follow up is the first outcome. The aim of the study is to highlight that the option early weight bearing (immediately in postoperative) is equal to the option delayed weight bearing.

ELIGIBILITY:
Inclusion Criteria:

* age: 40 to 65 years old
* patients with medial osteoarthritis of knee of level 1 or 2 from ahlback's classification with High Tibial Osteotomy indication
* one sided indication
* well understanding of information note by patient, non-opposition to perform the research
* Affiliation to a national health insurance program

Exclusion Criteria:

* age < 40 or > 65 years old
* medial osteoarthritis of knee of level superior to 2
* bilatéral indication
* patient opposition
* non affiliation to a national health insurance program
* law protected patients
* pregnancy and breast feeding

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-11; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
IKS score | one year follow-up

SECONDARY OUTCOMES:
IKS score | 6 months follow-up
VAS score of pain | at D1, D5, D15, M1, M2, M3, M6 and one year follow-up
IKDC (International Knee Documentation Committee) score | at M2, M, M6 and one year follow-up
Safety follow-up | during the one year follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Elvire SERVIEN, MD, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Result] Lansdaal JR, Mouton T, Wascher DC, Demey G, Lustig S, Neyret P, Servien E. Early weight bearing versus delayed weight bearing in medial opening wedge high tibial osteotomy: a randomized controlled trial. Knee Surg Sports Traumatol Arthrosc. 2017 Dec;25(12):3670-3678. doi: 10.1007/s00167-016-4225-8. Epub 2016 Jul 1. PMID 27371292